CLINICAL TRIAL: NCT00000689
Title: Phase I Trial of mBACOD and Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) in AIDS-Associated Large Cell, Immunoblastic, and Small Non-cleaved Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 074; 11048 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma, Non-Hodgkin; HIV Infections
Keywords: M-BACOD protocol; Nervous System Neoplasms; Infusions, Intravenous; Injections, Intravenous; Leucovorin; Cytarabine; Drug Evaluation; Drug Therapy, Combination; Granulocyte-Macrophage Colony-Stimulating Factor; Administration, Oral; Acquired Immunodeficiency Syndrome; Antineoplastic Agents, Combined
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; HIV Infections; Nervous System Neoplasms; Acquired Immunodeficiency Syndrome | interventions — Bleomycin; Vincristine; Doxorubicin; Cyclophosphamide; Methotrexate; Cytarabine; Leucovorin; sargramostim; Dexamethasone

INTERVENTIONS:
Drug: Bleomycin sulfate
Drug: Vincristine sulfate
Drug: Doxorubicin hydrochloride
Drug: Cyclophosphamide
Drug: Methotrexate
Drug: Cytarabine
Drug: Leucovorin calcium
Drug: Sargramostim
Drug: Dexamethasone

SUMMARY:
To determine the toxicity and effectiveness of adding sargramostim (recombinant granulocyte-macrophage colony stimulating factor; GM-CSF) to a standard chemotherapy drug combination (methotrexate, bleomycin, doxorubicin, cyclophosphamide, vincristine, and dexamethasone) known as mBACOD in the treatment of non-Hodgkin's lymphoma in patients who are infected with HIV.

Treatment of patients with AIDS-associated lymphoma is achieving inferior results when compared with outcomes for non-AIDS patients. Treatment with mBACOD has been promising, but the toxicity is very high. Patients treated with mBACOD have very low white blood cell counts. GM-CSF has increased the number of white blood cells in animal studies and preliminary human studies. It is hoped that including GM-CSF among the drugs given to lymphoma patients will prevent or lessen the decrease in white blood cells caused by mBACOD.

DETAILED DESCRIPTION:
Treatment of patients with AIDS-associated lymphoma is achieving inferior results when compared with outcomes for non-AIDS patients. Treatment with mBACOD has been promising, but the toxicity is very high. Patients treated with mBACOD have very low white blood cell counts. GM-CSF has increased the number of white blood cells in animal studies and preliminary human studies. It is hoped that including GM-CSF among the drugs given to lymphoma patients will prevent or lessen the decrease in white blood cells caused by mBACOD.

Patients admitted to the study receive chemotherapy in 21-day cycles. The length of therapy, 2 - 8 months, depends on how the tumor responds to treatment. Four medicines are given on day 1 of each cycle by vein (IV) (doxorubicin, cyclophosphamide, bleomycin, vincristine). Dosages of doxorubicin and cyclophosphamide are increased in later groups of patients if toxicity in the first group is tolerable. A fifth medicine (dexamethasone) is given by mouth (PO) on days 1 - 5 of each cycle and the sixth medicine (methotrexate) is given IV on day 15 of each cycle. Leucovorin is given after methotrexate to prevent methotrexate side effects. GM-CSF treatment is started on day 3 and continued for 11 days. To prevent the spread of the tumor, a spinal tap is done on 4 occasions to inject cytosine arabinoside directly into the spinal fluid. If tumor cells are present in the spinal fluid, the patient also takes cytosine arabinoside by spinal tap 3 x/week until the tumor cells disappear and then at monthly intervals for 1 year. Patients with tumor cells in the spinal fluid are also given radiation treatment to the head.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Positive HIV antibody by ELISA with Western blot confirmation, or positive HIV culture or serum p24 antigen capture assay, or prior diagnosis of AIDS by the CDC surveillance criteria.
* Pathological diagnosis of large cell (cleaved or non-cleaved), immunoblastic, or small non-cleaved lymphoma, stage I, II, III, or IV.
* If displaying systemic ("B") symptoms, evaluation for concurrent opportunistic infections as follows:
* Buffy coat for Mycobacterium intracellulare-avium (MAI) and cytomegalovirus (CMV) cultures; serum cryptococcal antigen; some measure of pulmonary function to exclude Pneumocystis carinii pneumonia including chest x-ray and either gallium scan, blood gases, or DLCO; stool culture and special stains for Salmonella, Isospora belli, cryptosporidium, CMV, and MAI in patients with diarrhea; computerized tomography (CT) scan or magnetic resonance imaging (MRI) of brain, or lumbar puncture for India ink, acid-fast bacilli smear, cryptococcal antigen, or fungal/mycobacterial culture.

Bone marrow involvement is permitted if the patient meets the hematologic criteria above.

Patients who have central nervous system (CNS) involvement at diagnosis or who are diagnosed during treatment will receive cranial radiotherapy:

- The total dose of 2400 rads will be delivered at a rate of 200 rads/day to the mid plane employing parallel opposing, lateral whole brain fields. The lower border of the field will encompass C2 to cover the meninges.

* Patients will be treated 5 days/week, Monday through Friday, until the total prescribed dose has been completed.
* Radiation will begin as soon as possible after documentation of lymphomatous disease in the CNS. If a second course of treatment is required, the 2400 rads is well within whole brain tolerance for normal tissues (4500-5000 rads).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Acute bacterial or opportunistic infection.
* Second primary cancer other than Kaposi's sarcoma, non-melanoma skin cancer, or carcinoma in-situ of the cervix.
* Primary central nervous system (CNS) lymphoma.

Concurrent Medication:

Excluded:

* Patients receiving prophylactic or maintenance therapy for bacterial or opportunistic infections, with the exception of those receiving Fansidar (sulfadoxine / pyrimethamine) for Pneumocystis carinii pneumonia prophylaxis.
* Antiretroviral agents.
* Immunomodulators.

Patients with the following are excluded:

* Acute bacterial or opportunistic infection.
* Second primary cancer other than Kaposi's sarcoma, non-melanoma skin cancer, or carcinoma in-situ of the cervix.
* Primary central nervous system (CNS) lymphoma.

Prior Medication:

Excluded:

* Prior therapy for lymphoma.
* Excluded within 1 week of study entry:
* Antiretroviral agents and immunomodulators.

Prior Treatment:

Excluded:

* Prior therapy for lymphoma.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18
Dates: Study Completion 1991-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walsh C, Study Chair; Levine AM, Study Chair
Locations (1):
- USC CRS, Los Angeles, California, United States

REFERENCES:
- [Background] Walsh C, Wernz JC, Levine A, Rarick M, Willson E, Melendez D, Bonnem E, Thompson J, Shelton B. Phase I trial of m-BACOD and granulocyte macrophage colony stimulating factor in HIV-associated non-Hodgkin's lymphoma. J Acquir Immune Defic Syndr (1988). 1993 Mar;6(3):265-71. PMID 7680712
- [Background] Redfield RR, Birx DL, Ketter N, Tramont E, Polonis V, Davis C, Brundage JF, Smith G, Johnson S, Fowler A, et al. A phase I evaluation of the safety and immunogenicity of vaccination with recombinant gp160 in patients with early human immunodeficiency virus infection. Military Medical Consortium for Applied Retroviral Research. N Engl J Med. 1991 Jun 13;324(24):1677-84. doi: 10.1056/NEJM199106133242401. PMID 1674589